CLINICAL TRIAL: NCT05156476
Title: Genicular Nerve Block Versus Femoral Triangle Nerve Block Versus LIA for Postoperative Analgesia After Total Knee Arthroplasty: A Pilot Randomized Controlled Superiority Trial
Brief Title: GENIFEM Trial: Postoperative Pain After Total Knee Arthroplasty (TKA)
Acronym: GENIFEM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Thibaut Vanneste, Principal Investigator, Ziekenhuis Oost-Limburg
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Z-2021085
Record Dates: First submitted 2021-09-20; First posted 2021-12-14 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Analgesia; Total Knee Arthroplasty
Keywords: Genicular block; iPACK; Local Infiltration Analgesia (LIA); Femoral triangle nerve block; Postoperative analgesia; Total knee arthroplasty
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Genicular nerve block-iPACK group (Active Comparator): Genicular nerve block-iPACK group (performed by anaesthesiologist) Method: Ultrasound and nerve stimulation guided injection Genicular nerve block will be performed on the the superomedial, the superolateral, the inferomedial and inferolateral genicular nerve.
  Drug: a total of 30 ml of ropivacaine 0.5% (150 mg) will be used for this treatment arm.
  Interventions: Procedure: Genicular nerve block-iPACK group
- Femoral triangle block-iPACK group (Active Comparator): Femoral triangle block-iPACK group (performed by anaesthesiologist) Method: Ultrasound and nerve stimulation guided injection Drug: a total of 30 ml of ropivacaine 0.5% (150 mg) will be used for this treatment arm
  Interventions: Procedure: Femoral triangle block-iPACK group
- Local Infiltration Analgesia (LIA) (Active Comparator): LIA (performed by surgeon) Method: Blind injection Drug: a total of 200 ml of 0.2% ropivacaine will be used (400 mg). Of this, 150 ml of ropivacaine 0.2% will be mixed with 1 mg of adrenaline.
  Interventions: Procedure: Local infiltration analgesia

INTERVENTIONS:
Procedure: Genicular nerve block-iPACK group — Group 1: Genicular nerve block-iPACK group (performed by anaesthesiologist) Method: Ultrasound and nerve stimulation guided injection Drug: a total of 30 ml of ropivacaine 0,5% (150 mg) will be used
  Arms: Genicular nerve block-iPACK group
Procedure: Femoral triangle block-iPACK group — Group 2: Femoral triangle block-iPACK group (performed by anaesthesiologist) Method: Ultrasound and nerve stimulation guided injection Drug: a total of 30 ml of ropivacaine 0,5% (150 mg) will be used
  Arms: Femoral triangle block-iPACK group
Procedure: Local infiltration analgesia — Group 3: LIA (performed by surgeon) Method: Blind injection Drug: a total of 200ml of 0.2% ropivacaine will be used (400mg). Of this, 150ml of ropivacaine 0.2% will be mixed with 1mg of adrenaline.
  Arms: Local Infiltration Analgesia (LIA)

SUMMARY:
Motor-sparing analgesic interventions for patients undergoing total knee arthroplasty (TKA) are a key component of fast-track surgery.

The investigators want to estimate treatments effects, inclusion rate, and feasibility of conducting a future randomized controlled superiority trial and to assess whether the short-term postoperative analgesic effect and ambulation after a Genicular - Infiltration Between Popliteal Artery and Capsule of Knee (iPACK) block in patients undergoing unilateral primary TKA is superior to Femoral triangle - iPACK block and Local Infiltration Analgesia (LIA).

The study is a prospective, double-blind, triple-arm superiority pilot randomised controlled trial with a randomization rate 1:1:1.Group I will receive a Genicular - iPACK block, group II a Femoral Triangle - iPACK block and group III LIA.

The primary study outcome is the proportion of patients that are able to mobilise (defined as walk 10 meters with assistance) with a numerical rating scale (NRS) of equal or less than 4 without the use of opioids at 4-6 hours after TKA. Secondary outcomes are efficacy (measured in NRS, total morphine consumption, total morphine titrations), functionality (quadriceps strength, timed-up-and-go, 6-minute walk test, inpatient falls), frequency of opioid related adverse events, discharge readiness, patient satisfaction, health-related quality of life, length of stay (LOS), complications after TKA and adverse events related to the study interventions.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is one of the most frequently performed orthopedic surgical procedures for the treatment of osteoarthritis of the knee. Fast-tract recovery protocols emphasize the importance of early mobilization and physiotherapy to improve functional recovery, reduce postoperative complications, and decrease the economic burden of TKA. As the patients having TKA typically have severe pain postoperatively, multimodal analgesic regimen in many institutions includes interventional analgesia modality, such as nerve blocks, to facilitate early mobilization. At this time however, no universal recommendation exists on what constitutes the optimal nerve block technique that provides favorable balance between motor sparing for ambulation and analgesia.

Various motor-sparing nerve blocks (e.g., femoral triangle block, adductor canal block, obturator nerve blocks, Infiltration Between Popliteal Artery and Capsule of Knee (iPACK), genicular nerve block and Local Infiltration Analgesia (LIA)) are viable options for interventional analgesia in patients undergoing TKA. By this study in patients having TKA, the investigators aim to compare the analgesia and ambulation between the genicular nerve block iPACK versus Femoral triangle nerve block + iPACK versus LIA.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age at screening
* Scheduled to undergo elective primary unilateral TKA
* American Society of Anaesthesiologists (ASA) physical status 1, 2 or 3
* Mentally competent to provide informed consent, to report pain intensity and to use patient-controlled analgesia
* Physically able to perform independently the baseline functionality tests

Exclusion Criteria:

* Obesity (BMI>40)
* Previous open knee surgery
* Revision TKA or bilateral TKA
* Contraindication to the following study medication: ropivacaine, morphine, midazolam, ketorolac, propofol, remifentanil, clonidine, dexamethasone, acetaminophen
* Uncontrolled anxiety, psychiatric, or neurological disorder that might interfere with study assessments
* Chronic widespread pain
* Radicular pain in index legClinical Study Protocol Version 1.0
* Preoperative strong opioid use within 3 days before surgery (with the exception of weak opioids: tramadol and codeine)
* Any chronic neuromuscular deficit affecting the peripheral nerves or muscles of the surgical extremity
* Impaired kidney function (Chronic kidney disease (CKD) G4-G5 according to Kidney Disease: Improving Global Outcomes (KDIGO) classification)
* Alcohol or drug abuse
* Pregnant, nursing or planning to become pregnant before treatment. Women of reproductive age will be tested on pregnancy prior to start of the study. Participants who get pregnant after the treatment during the follow-up period will not be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
Pain assessed by NRS at rest and movement: 4 -6 hours after TKA | 4 to 6 hours after TKA
  The main study outcome is the proportion of patients that have a numeral rating scale (NRS) <4 during mobilization without morphine at 4-6 hours after TKA. Mobilisation will be defined as walking 10 meters with walking aids or an assistant. NRS is a unidimensional, subjective measurement of pain intensity, expressed by the patient as a number between 0 and 10. It is a 11 point scale in which 0 equals no pain and 10 maximal pain. NRS at rest will also be determined

SECONDARY OUTCOMES:
Pain assessed by NRS | 24 hours, 48 hours, 72 hours and 1 month
  NRS is determined at rest and movement at 24 hours, 48 hours, 72 hours and 1 month after TKA. NRS is a unidimensional, subjective measurement of pain intensity, expressed by the patient as a number between 0 and 10. It is a 11 point scale in which 0 equals no pain and 10 maximal pain.
Post-operative morphine consumption and titration | 4-6 hours, 24 hours, 48 hours and 72 hours after TKA
  The amount of morphine that the patient demanded and that was given will be determined at 4-6 hours, 24 hours, 48 hours and 72 hours after TKA
Quadriceps strength pre-and post operative | baseline, 4-6 hours, 24 hours, and 48 hours after TKA
  quadriceps strength measured in maximum voluntary isometric contraction (MVIC) at baseline (pre-operative), 4-6 hours, 24 hours, 48 hours after TKA
6-minute walking test pre-and post operative | baseline, 24 hours, 48 hours and 72 hours after TKA
  The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity. The 6 minute walking test will be performed at baseline (pre-operative), 24 hours, 48 hours and 72 hours after TKA
Timed up and go pre- and post operative | baseline, 24 hours, 48 hours and 72 hours after TKA
  In the timed up and go test, subjects are asked to rise from a standard armchair, walk to a marker 3 m away, turn, walk back, and sit down again. The results are expressed in minutes or seconds. The timed up and go test will be performed at baseline (pre-operative), 24 hours, 48 hours and 72 hours after TKA
Health status assessed by WOMAC: pre- and post-operative | baseline and 1 month after TKA
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is a widely used self-administered health status measure used in assessing pain, stiffness, and function in patients with osteoarthritis of the knee.
  The test questions are scored on a scale of 0-4. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations. The questionnaire will be performed at baseline (pre-operative) and 1 month after TKA
The change in health-related quality of life assessed by EuroQol-5 Dimension-5 Level (EQ-5D-5L) questionnaire | baseline and 1 month after TKA
  The EQ-5D-5L is a patient-reported generic measure of HRQoL comprising five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Responses to the 5 items (one for each dimension) result in a patient's health state that can be transformed into a utility score ranging between 0 (death) and 1 (full health), representing the quality of life of the health state.
Assessment of anxiety and depression by the Hospital Anxiety and Depression Scale (HADS) questionnaire | baseline and 1 month after TKA
  HADS is developed to detect anxiety and depression in patients with physical health problems. The questionnaire consists of 14 items: 7 items to measure anxiety and 7 items to measure depression
Measurement of patient satisfaction by the patient satisfaction scale | 72 hours and 1 month after TKA
  The patient satisfaction scale is measured in a 5-point Likert scale with response categories consisting of very satisfied, somewhat satisfied, neutral, somewhat dissatisfied, and very dissatisfied
Assessment of pain experience by the Pain Catastrophizing Scale (PCS) | baseline and 1 month after TKA
  The PCS is often used in clinical settings to measure catastrophic thinking related to pain. The 13 item questionnaire consists of 3 subscales (magnification, rumination and helplessness) and asks patients to reflect on past painful experiences and to indicate the degree on which they experiences each of 13 thoughts of feelings on a 5- point scale (0 not at all and 4 all the time).
Nerve block time | per-operative
  (time from first needle insertion to final needle exit)
Number and type of complications of TKA | Through study completion, up to 1 month after randomisation and study intervention
  Complications of TKA (e.g., transfusions, prevalence of venous thrombo-embolic event, infection…) will be assessed per - and post-operative
Discharge readiness | Through study completion, up to 1 month after randomisation
  The discharge readiness will be compared between the three groups.
  Discharge readiness is assessed by means of the following:
  * Pain is under control (<4) with oral painkillers
  * Wound is dry (not purulent)
  * Knee flexion is possible over 70 degrees
  * Patients are self-sustainable with crutches
  The discharge readiness is described as yes or no.
Length of stay | Through study completion, up to 1 month after randomisation
  The length of stay will be compared between the three groups by counting the number of days in the hospital
Number of hospital readmissions (due to knee related problems at 1 month) | 1 month after TKA
  The readmission status of patients will be compared between groups after 1 month of TKA.
Safety assessment by reporting adverse events | Through study completion, up to 1 month after randomisation
  Throughout the study, adverse events related to the intervention will be collected.
Frequency of opioid related adverse event | 0 hours, 4-6 hours, 24 hours, 48 hours and 72 hours after TKA
  The frequency of opioid related adverse event will be assessed from the start of surgery until 72 hours after TKA
Attributable mortality during the trial | during hospitalisation, an average of 3 days
  Mortality which is attributable to study interventions, surgical procedure, underlying condition or other relevant reasons will be investigated during the trial (perioperative, until discharge)
Inpatient fall | during hospitalisation, an average of 3 days
  The risk of inpatient fall will be assessed during hospital stay.

OTHER OUTCOMES:
Success of blinding | 72 hours after TKA
  Patients will be asked to guess their treatment allocation at 72 hours after TKA

CONTACTS AND LOCATIONS:
Overall Officials: Thibaut Vanneste, MD, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium

REFERENCES:
- [Derived] Belba A, Peene L, Mesotten D, Vanlommel L, Van Zundert J, Vanneste T; Collaborators. The GENIFEM Pilot Randomized Trial: Genicular Nerve Block vs Femoral Triangle Block vs Local Infiltration Analgesia for Total Knee Arthroplasty. Anesth Analg. 2026 Jan 1;142(1):186-189. doi: 10.1213/ANE.0000000000007622. Epub 2025 Jul 3. No abstract available. PMID 40608549